CLINICAL TRIAL: NCT06758024
Title: Multicentric Evaluation of a Strategy for Early Infliximab Optimization Among Adult Inflammatory Bowel Disease Patients
Brief Title: PROactive and Early Infliximab Monitoring and OPTimization in Inflammatory Bowel Disease
Acronym: PROMPT-IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Clínica Universidad de los Andes (Other); Hospital San Juan de Dios,Chile (Other); University of Chile (Other); Clinica Indisa (Other); Universidad de La Frontera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240320009; SA24I0002 (Other Grant/Funding Number: The Chilean National Research and Development Agency (ANID))
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: Inflammatory Bowel Disease; Infliximab; dashboard-guided dosing; therapeutic drug monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Multicenter Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dashboad-guided dosing (Other): Eligible patients will receive IFX with proactive therapeutic drug monitoring during induction (week 2 and 6) and dashboard-guided dosing options will be suggested to their attending gastroenterologists
  Interventions: Drug: Infliximab
- Standard dosing (Other): Eligible patients will receive IFX standard dosing during induction based solely on clinical data
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — IFX therapeutic drug monitoring before the second and third infusion and subsequent dashboard-guided dosing regimes suggested to attending gastroenterologists based on clinical and pharmacokinetics data
  Arms: Dashboad-guided dosing
Drug: Infliximab — No IFX therapeutic drug monitoring before the second and third infusion and subsequent dosing regimes based on clinical data
  Arms: Standard dosing

SUMMARY:
Infliximab (IFX) is a Food and Drug administration (FDA)-appoved monoclonal antibody medication targeting tumor necrosis factor (TNF) widely used in inflammatory bowel disease (IBD) to treat intestinal inflammation and improve patient's symptoms. Intravenous (iv) IFX is effective to treat hospitalized IBD patients with moderate-to-severe flares who fail iv corticosteroids (CS). However, about one-third of IBD patients do not respond to this medications and a half will loss the response after an initial response. Researchers have shown that most of these phenomena occur due to low IFX concentrations sometimes accompanied by the development of anti-drug antiboides (ADA) againts IFX.

Blood concentrations of IFX are widely variable among IBD patients despite receiving the same weight-based dose. Several patient factors including laboratory parameters and severity of intestinal inflammation influence the way an individual's body proccesses and eliminate this type of medications. Dashboard software systems can take into account patient characteristics and IFX concentrations to modelate and facilitate dosing of IFX. By using pharmacokinetics (PK) models specifically developed to facilitate IFX dosing, these softwares can provide and recommend multiple dosing regimes to help the clinicians to select the appropriate dose to achieve target and optimal IFX concentrations.

The goal of this clinical trial is to learn if early measuring of IFX blood concentrations and dashboard-guided IFX dose adjustment in Chilean IBD patients starting IFX, increases the proportion of patients with optimal IFX levels and improves patient outcomes. Researchers will measure IFX concentrations before the second (week 2) and third dose (week 6) in a prospectively collected individual patient cohort and this information along with clinical data will be analyzed with a dashboard software system and multiple dosing regime options will be provide to the attending clinicians to facilitate the selection of the next IFX weight-based dose and interval of infusions. This group will be compared with IBD patients with standard of dosing where attending clinicians make the dosing decisions based on clinical parameters. The main goal is to analyze if IBD patients in the dashboard-guided dosing arm achieve a higher proportion of optimal IFX concentrations at week 14 of treatment, develop ADA less frequently and improve clinical outcomes compared with standard dosing group.

Participants will be asked to:

* Provide clinical data about their disease and other conditions
* Provide blood samples at enrollment and before each IFX infusion (IFN) during one year
* Maintain regular clinical assessments every 3 months for one year

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are chronic diseases that entail important morbidity and frequently require high-cost medications such as biologic therapies. Monoclonal antibodies against tumoral necrosis factor (anti-TNF) are effective and can modify the progressive course of IBD. In Chile, given the high cost of anti-TNF therapy, this medication is provided by a national program with universal coverage. Unfortunately, a significant proportion of IBD patients never respond (primary non-response, PNR) or experience loss of response (secondary loss of response, SLR) to anti-TNF within the first year of therapy and current evidence support that the complex pharmacokinetics of anti-TNF is involved in both scenarios. Additionally, low trough levels (TL) are associated with the development of antidrug antibodies (ADA) which reduce anti-TNF efficacy and can cause anaphylactic reactions. This is particularly relevant for intravenous infliximab (IFX) which is usually indicated in IBD patients with acute severe disease not responding to iv corticosteroids. Therefore, IFX is frequently dose escalated in patients based on clinical parameters that are thought to be related to drug clearance with conflicting evidence supporting this strategy. Several studies have demonstrated that IFX TL between 7-20 mcg/ml at week 14 of treatment is a strong and independent predictor of therapy response. Furthermore, IFX dashboard-guided dose optimization based on clinical and pharmacokinetic (PK) parameters using adaptive Bayesian modeling have demonstrated to be more precise that empirical adjustments based on the clinician intuition alone. Therefore, the goal of this study is to analyze whether early therapeutic drug monitoring (TDM) and dose adjustment based on a Bayesian model (iDOSE) in CD and UC patients initiating IFX, increases the proportion of patients with therapeutic levels (7-20 mcg/ml), reducing immunogenicity and consequently increasing the rate of disease remission. A prospective multicentric randomized clinical trial (RCT) of Chilean adult IBD inpatients starting IFX due to moderate-to-severe disease refractory to corticosteroids will be carried out. Patients will be randomized 1:1 to:

1. - Dashboard-guided dosing arm. Patients will undergo proactive TDM during induction (TL at IFN 2 and 3) with dose adjustment based on iDOSE.
2. - Standard dosing arm. Patients will receive dose adjustment based solely on clinical parameters.

Both groups will be followed-up after induction with clinical visits, TL and ADA at week 14 (INF 4), 26 and 52. Researchers expect that a higher proportion of patients in the dashboard-guided dosing arm will achieve therapeutic TL of IFX (7-20 mcg/ml) at week 14 of treatment (Primary outome). Secondary outcomes will include clinical and laboratory parameters related to therapy response at week 52 of treatment, proportion of patients experiencing PNR and SLR, patients developing ADA, as well as, adverse events, hospitalization and surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients with Crohn's disease, ulcerative colitis or inflammatory bowel disease-unclassified.
* Moderate-to-severe flare who fail to iv steroids and require infliximab as per standard of care by treating gastroenterologist

Exclusion Criteria:

* Participant younger than 18 years
* Non-controlled infectious diseases
* Permanent ileostomy or Ileal pouch-anal anastomosis
* Pregnancy
* Patients do not consent to participate in study
* Patients unable to comply with protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Infliximab optimal concentration | Week 14
  Proportion of patients who achieve infliximab trough levels between 7-20 mcg/ml at week 14 of treatment

SECONDARY OUTCOMES:
Clinical remission | Week 52
  Proportion of subjects in clinical remission at week 52 (CDAI <150 for CD or partial Mayo score < 2 for UC).
Corticosteroid-free clinical remission | Week 52
  Proportion of subjects in Corticosteroid (CS)-free clinical remission at week 52 (CDAI <150 for CD or partial Mayo score < 2 for UC and no use of CS within previous 6 months).
Sustained corticosteroid-free clinical remission | Week 52
  Proportion of subjects with sustained CS-free clinical remission at week 52 (CDAI <150 for CD or partial Mayo score < 2 for UC and no CS use from week 14 through week 52).
CRP normalization | Week 52
  Proportion of subjects with normalisation of C-reactive protein (CRP) at week 52 (decrease from ≥1 at baseline to <1 mg/dL).
Fecal calprotectin normalization | Week 52
  Proportion of subjects with normalisation of fecal calprotectin at week 52 (decrease from >250μg/g at baseline to ≤250mcg/g).
Primary non-response | Week 14
  Proportion of subjects who are primary non-responders (≤70-point decrease in CDAI score for CD or decrease in partial Mayo score of ≥2 points and ≥25% for UC from baseline) and at least one of: CRP ≥1mg/dL or FC >250μg/g; or need for rescue therapy prior to week 14).
Secondary loss of response | Week 14 through 52
  Proportion of subjects exhibiting secondary loss of response (CDAI >220 or partial Mayo score >4 and at least one of: CRP ≥1mg/dL or FC >250μg/g; or need for rescue therapy) during maintenance.
Antibodies to infliximab-free survival | Week 2 through 52
  Proportion of subjects with no antibodies to infliximab (ATI).
Proportion of subjetcs with antibodies to infliximab | Week 2 through 52
  Proportion of subjects with antibodies to infliximab (ATI)
Time to antibodies to infliximab | Week 2 through 52
  Time to antibodies to infliximab (ATI) development.
Adverse events | Week 0 through 52
  Proportion of subjects with any treatment-related adverse event.
Surgery | Week 0 through 52
  Proportion of subjects with CD or UC-related surgery
Time to surgery | Week 0 through 52
  Time to CD or UC-related surgery
Hospitalization | Week 0 through 52
  Proportion of subjects with CD or UC-related hospitalisation.
Time to hospitalization | Week 0 through 52
  Time to CD or UC-related hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Catolica of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided